CLINICAL TRIAL: NCT05233592
Title: Glycemic Effects of the COVID-19 Booster Vaccine in Type 1 Diabetes
Status: Completed | Type: Observational
Sponsor: Johns Hopkins University (Other)
Collaborators: DexCom, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: IRB00305567
Record Dates: First submitted 2022-02-09; First posted 2022-02-10 (Actual); Last update posted 2023-05-17 (Actual); Status verified 2023-05

CONDITIONS: Type 1 Diabetes; Diabetes Mellitus, Type 1
Keywords: COVID-19; Vaccine; Hyperglycemia; Insulin Resistance; Continuous Glucose Monitor; CGM; Booster
MeSH Terms: conditions — Diabetes Mellitus, Type 1; COVID-19; Hyperglycemia; Insulin Resistance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- T1D Patients Using CGM: Type 1 Diabetes patients using CGM who have received COVID-19 vaccine booster shot (first or second)
  Interventions: Device: CGM

INTERVENTIONS:
Device: CGM — Patients wear a CGM to measure the effects of the COVID-19 booster vaccine on blood sugar levels.

SUMMARY:
Vaccines for COVID-19 are an essential part of combating the coronavirus pandemic. Vaccines "prime" the immune system against an invader (in this case the SARS-CoV-2 virus) by causing a temporary increased immune or inflammatory response. Inflammation can temporarily increase sugar levels and/or insulin requirements among patients with diabetes. The purpose of this study is to investigate whether the "booster" COVID-19 vaccine dose causes temporarily increased sugar levels and/or insulin dose requirements among patients with Type 1 Diabetes (T1D).

DETAILED DESCRIPTION:
Over 30 million people in the US have diabetes. It's well known that acute inflammation can temporarily increase blood sugar levels (hyperglycemia) and insulin resistance among patients with diabetes, particularly those with type 1 diabetes (T1D). Vaccines cause an inflammatory reaction, because the vaccines prime the body's immune system against a potential virus. Reports have described temporary hyperglycemia and/or insulin resistance after COVID vaccine administration. However, to date this has not been studied in a rigorous fashion. The objective of the study is to determine if the COVID-19 booster causes increased sugar levels and insulin dose adjustments in patients with T1D. This is a study in adult patients with Type 1 Diabetes who have not yet received the COVID-19 booster vaccine. The study consists of two short outpatient (clinic) visits. Visit 1 occurs 3-5 days before receiving the COVID-19 booster vaccine (pre-vaccine visit). During this visit, the participant will fill out a questionnaire and have a blinded Dexcom G6 Pro CGM applied to the participant. An optional second "backup" Dexcom G6 Pro CGM will be provided, in case the first continuous glucose monitor (CGM) falls off accidentally. Visit 2 occurs 10 days after Visit 1 (about 5 days after receiving the first or second booster vaccine shot), at which time the CGM would be removed. Participants will continue participants' usual routine diabetes care while participating in the study, including using the participants' own glucometer or CGM. Participants will also be asked to keep track of participants' insulin doses administered during the 10-day study.

ELIGIBILITY:
Inclusion Criteria:

1. Adult (age ≥18yo)
2. Type 1 Diabetes
3. Is already fully vaccinated against COVID-19 (e.g. received 2 doses of Pfizer or Moderna or one dose of Johnson & Johnson)
4. Available to receive a COVID-19 booster vaccine (first or second booster dose)

Exclusion Criteria:

1. Has already received a COVID-19 booster vaccine dose
2. Known physical or psychological disorder which would prohibit the patient from complying with the study procedures (e.g. allergy to adhesive, profound skin disorder, known to have severe adverse reactions previously to CGMs, poorly controlled schizophrenia, etc.)
3. Recent, acute, or chronic medical condition which may significantly affect insulin resistance or measurements of glucose (e.g. severe cirrhosis, acute infection, cancer on chemotherapy, etc.)
4. On a medication known to cause significant hyperglycemia (e.g. supraphysiologic dose of steroids) or negatively affect readings of CGM (e.g. supraphysiologic doses of acetaminophen (e.g. >4g/d)).
5. Pregnant or actively trying to get pregnant
6. Planned PET, CT, or MRI test in the next 10 days
7. Unwilling or unable to keep track of insulin usage during the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with Type 1 Diabetes who have received either 2 doses of Moderna/Pfizer COVID-19 vaccine or 1 dose of Johnson & Johnson, but have not yet received their COVID-19 booster (first or second booster dose).
Sampling Method: Non-Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2022-03-08 (Actual); Primary Completion 2023-04-04 (Actual); Study Completion 2023-04-04 (Actual)

PRIMARY OUTCOMES:
Total Daily Insulin Resistance (TDIR) | Day 1 post-vaccine as compared to baseline
  Mean glucose multiplied by total daily insulin dose.

SECONDARY OUTCOMES:
Change in TDIR | Days 1 to 5 post-vaccine as compared to baseline
  Mean glucose multiplied by total daily insulin dose.
Change in Time in Range | Day 1 post-vaccine as compared to baseline
  Percentage of time that the participant's blood sugar is between 70-180mg/dL.
Change in Daily Insulin Requirement | Day 1 post-vaccine as compared to baseline
  Total Daily insulin dose.
Change in Time in Hyperglycemia | Day 1 post-vaccine as compared to baseline
  Percentage of time that participants' sugar level is above 180mg/dL.

OTHER OUTCOMES:
Post-hoc ANOVA | Days 1 to 5 post-vaccine as compared to baseline
  One-way Repeated Measures ANOVA will be used to assess changes in secondary outcome variables over time.
Post-hoc t-test | Days 1 to 5 post-vaccine as compared to baseline
  Assess whether secondary variables from individual days are significantly different from baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew P Demidowich, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Cardiovascular Specialists of Central Maryland, Columbia, Maryland, United States